CLINICAL TRIAL: NCT05682287
Title: The Effect of Capacitive and Resistive Monopolar Radiofrequency of 448 kHz on Pain and Function in People Diagnosed With Lumbar Pain Syndrome
Brief Title: The Effect of Radiofrequency of 448 kHz on Pain and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Health Sciences (Other)
Responsible Party: Principal Investigator, Ivan Jurak, Head of Physiotherapy, University of Applied Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 602-04/21-25/840
Record Dates: First submitted 2022-12-24; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Chronic Low-back Pain; Lumbago; Low Back Pain, Recurrent
Keywords: chronic low back pain; 448kHz capacitive resistive monopolar radiofrequency; randomised controlled trial; pain; disability
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants in the experimental group will be treated with a combination of 448kHz capacitive resistive monopolar radiofrequency and Proprioceptive neuromuscular facilitation (PNF) over the course of two weeks.
  1. 448 kHz radio frequency therapy will be carried for a duration of 15 min. Contact cream will be applied beforehand to increase the electrical conductivity in the treated area.
  2. After the radiofrequency therapy, participants will exercise for exactly 20 minutes using the PNF concept exercises to mobilize the pelvis and lumbar spine, primarily strengthening the muscles of the abdomen, back and hips.
  Therapy will be administered for a total of 5 times in two weeks. Three times in week 1 and two times in week 2.
  Interventions: Device: 448kHz capacitive resistive monopolar radiofrequency; Other: Proprioceptive Neuromuscular Facilitation
- Control group (Active Comparator): Participants will exercise for exactly 20 minutes, over the course of two weeks, using the PNF concept exercises to mobilize the pelvis and lumbar spine, primarily strengthening the muscles of the abdomen, back and hips.
  Therapy will be administered for a total of 5 times in two weeks. Three times in week 1 and two times in week 2.
  This is identical intervention and the second intervention in the experimental group.
  Interventions: Other: Proprioceptive Neuromuscular Facilitation

INTERVENTIONS:
Device: 448kHz capacitive resistive monopolar radiofrequency — Capacitive resistive monopolar radiofrequency (CRM) treatment is a type of medical procedure that uses radiofrequency energy to heat the targeted tissue.
  Arms: Experimental group
Other: Proprioceptive Neuromuscular Facilitation — Proprioceptive neuromuscular facilitation (PNF) is a type of physical therapy that uses techniques such as stretching and strengthening exercises to improve muscle function and movement patterns.
  Other Names: PNF

SUMMARY:
The goal of this trial is to compare the effects 448kHz capacitive resistive monopolar radiofrequency (CRM) with Proprioceptive Neuromuscular Facilitation (PNF) versus only PNF in chronic low back pain patients.

The main questions it aims to answer are:

1. Is there any difference in interventions on reduction of pain.
2. Is there any difference in interventions on reduction of disability.

Participants will in the experimental group will be treated with a combination of:

1. 448kHz capacitive resistive monopolar radiofrequency and,
2. PNF intervention

Participants will in the control group will be treated only using

1. PNF intervention (identical to experimental group)

Researchers will compare experimental and control group to see if there are differences in reduction of pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years, chronic low back pain (CLBP)

Exclusion Criteria:

* spinal fractures, radiculopathies, history of spinal surgery, spinal stenosis, history of thrombosis, pacemaker, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline: Pain - Visual Analogue Scale (VAS) | Change from baseline pain after two weeks (14 days).
  Change from baseline pain, measured by 0-10 Visual Analogue Scale (VAS). VAS has a minimum score of 0 and a maximum score of 10. Higher score indicates a worse outcome (e.g., greater pain intensity).
Change from baseline: Disability - ODI (Oswestry Low Back Pain Disability Questionnaire) | Change from baseline disability after two weeks (14 days).
  Change from baseline disability, measured by Oswestry Low Back Pain Disability Questionnaire. ODI has a minimum score of 0% and maximum score of 100%. Higher score indicates a worse outcome (e.g., greater disability).

SECONDARY OUTCOMES:
Change from baseline: Disability - Quebec Back Pain Disability Scale (QBPD) | Change from baseline disability after two weeks (14 days).
  Change from baseline disability, measured by Quebec Back Pain Disability Scale. QBPD has a minimum score of 20 and maximum score of 100. Higher score indicates a worse outcome (e.g., greater disability).
Change from baseline: Roland-Morris Disability Questionnaire (RMDQ) | Change from baseline disability after two weeks (14 days).
  Change from baseline disability, measured by Roland-Morris Disability Questionnaire. RMDQ has a minimum score of 0 and maximum score of 24. Higher score indicates a worse outcome (e.g., greater pain-related disability).

CONTACTS AND LOCATIONS:
Locations (1):
- Polyclinic Cerebellum, Varaždin, Varaždin County, Croatia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized IPD will be shared either as a supplement to manuscript or on adequate server for storing IPD data.
  Data will always be available upon inquiry by email to lead investigators. All variables that were measured will be included in the dataset.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When: Upon publication. How long: Indefinitely.
Access Criteria: Available to all. No criteria for accessing the data.

REFERENCES:
- [Derived] Jurak I, Grabar S, Zura N, Jakus L. Evaluating the Efficacy of Capacitive Resistive Monopolar Radiofrequency Combined With Proprioceptive Neuromuscular Facilitation in Managing Chronic Low Back Pain: A Randomised Controlled Trial. Physiother Res Int. 2025 Jan;30(1):e70009. doi: 10.1002/pri.70009. PMID 39572389